CLINICAL TRIAL: NCT06394271
Title: WARRIORS Trial and Registry
Brief Title: Early Endovascular Repair Versus Surveillance for Women With Small Abdominal Aortic Aneurysm
Acronym: WARRIORS
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Imperial College London (Other)
Collaborators: University College, London (Other); University of Leicester (Other); St Georges University Hospital (Unknown); University of Southern Denmark (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: 24CX8836
Record Dates: First submitted 2024-04-19; First posted 2024-05-01 (Actual); Last update posted 2025-03-20 (Actual); Status verified 2025-03

CONDITIONS: Abdominal Aortic Aneurysm
Keywords: abdominal aortic aneurysm; women's health; intervention threshold; endovascular aneurysm repair
MeSH Terms: conditions — Aortic Aneurysm, Abdominal

STUDY DESIGN:
Intervention Model Description: Women will be randomised 1:! to either early endovascular aneurysm repair or to routine surveillance until the aneurysm diameter reaches 5.5 cm. Randomisation will be stratified by country, age ( below 76 years or older) and aneurysm diameter (4.0-4.9 cm and larger).
Who Masked: Outcomes Assessor
Masking Description: Endpoint adjudication committee will be blinded to randomisation allocation.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Early EVAR (Experimental): Endovascular aneurysm repair within 2 months of randomisation using any licensed infrarenal aortic endograft within the manufacturer's instructions for use.
  Interventions: Device: EVAR
- Surveillance (No Intervention): Regular imaging surveillance (ultrasound or CT) of aneurysm diameter until the diameter reaches 5.5 cm, develops symptoms of impending rupture or ruptures. The delayed repair may be by any method.

INTERVENTIONS:
Device: EVAR — Catheter based insertion of aortic endograft via iliac or femoral arteries
  Other Names: infrarenal aortic endograft
  Arms: Early EVAR

SUMMARY:
Elective Abdominal Aortic Aneurysm (AAA) repair is offered when the risk of rupture exceeds the risk of surgery. Women (versus men) have a four-fold higher risk of AAA rupture but almost double the operative mortality. It is unknown whether the current 5.5cm diameter AAA repair threshold, derived from randomised trials including only 4% women, is applicable to women.

Therefore, should women have their aneurysms repaired electively at smaller diameters than men to improve their AAA-related survival and quality of life? WARRIORS is an international randomised controlled trial of early elective endovascular repair versus routine surveillance in women (n=1112) with small asymptomatic AAA (4-5.4cm diameter), nested within a registry of non-participants. The surveillance group will be offered repair for rupture or upon reaching the 5.5cm threshold. Randomisation will be 1:1 stratified by country, age, and aneurysm diameter. The trial is powered for aneurysm-related mortality or rupture at 5 years. Quality-Adjusted-Life-Years is a major secondary outcome. Other outcomes include: operative mortality and complications, anxiety, major cardiovascular adverse events, and cost-effectiveness. Quality-of-life and anxiety questionnaires and "standard-of-care" using routine data will be collected.

The trial aims to progress health equity through provision of evidence for sex-specific clinical guidelines for AAA repair.

DETAILED DESCRIPTION:
Design

WARRIORS (Women's Aneurysm Research: Repair Immediately Or Routine Surveillance) is an international, multicenter, open label, superiority RCT, randomly allocating consenting with small abdominal aortic aneirysm (AAA), morphologically eligible for endovascular repair (EVAR), in a 1:1 ratio to either early AAA repair by EVAR or to routine ultrasonographic surveillance. It will have a Vanguard phase with adjudicated endpoints. Each participant will be followed up for 5-years.

It is planned that the UK will provide13.5%of total target recruitment. The remaining patients will be recruited in mainland Europe (32.5% North America and Australasia (4.5%)

The trial will start with an international Vanguard phase of 250 patients,, to optimise and confirm randomization rates and patient safety (operative mortality rate) and ensure inclusivity of underserved groups. In both the UK and other countries, the Vanguard phase is scheduled to start in April 2025. Women will be recruited over 12 months during which period there will be an ongoing programme of qualitative research to optimise recruitment and ensure representation of minority and underserved groups. The Vanguard trial will run for a further 6 months, to allow completion of interventions and post-operative follow up and analysis of the results. The international Vanguard trial is scheduled to run for one year following the opening of >25% of target sites per participating country to assess and feasibility (recruitment) and safety (operative mortality, aneurysm exclusion and complications). support recruitment rates. The Vanguard phase should be completed within the first 30- months of the trial and include a total of 250 women (including 50 from the UK) and with total accrual of 35 patients/month between months 6-12. The qualitative work to optimise recruitment will use the Quintet Recruitment Intervention (QRI) [12], to identify recruitment obstacles and facilitate improvements to the recruitment process, and the SEAR framework [13], to capture ethnic and diversity characteristics and highlight any discrepancies in the recruitment process, which may negatively impact underserved groups participating (details given below). If only 150-249 have been recruited, improvement measures/additional centres will be introduced to achieve the target accrual of 35/month, with re-evaluation (after a further 6 months). Remedial measures could include visiting and motivating centers, implementation of actions arising from the qualitative work (including improving patient-facing material), running focus groups with those identifying patients including vascular nurses and sonographers, the opening of reserve sites, and an incentive programme (e.g. rewards for recruiting every 50th or 1100th woman). If <150 patients have been randomised and current monthly recruitment is <35/month for months 10-12, the trial should be stopped.

The results of the Vanguard trial should enable the Data Monitoring and Ethical Committee (DMEC) to set stopping rules for the rest of the trial, based on operative mortality and major complications. In the Vanguard phase, we propose that 30-day mortality for early elective EVAR group should not exceed 3%, but this will need the agreement of the DMEC.

The performance and results of the Vanguard trial will be scrutinized by both the Trial Steering Committee and the DMEC.

Identification and recruitment of participants

Women with small AAA, 4.0-5.4 cm (based on local measurements by ultrasound) being monitored for AAA growth in hospital or community screening and surveillance programmes. Women also may be identified from imaging studies for other conditions, with referral to vascular surgeons, in which case the CT or other imaging measurement 9centre line orthogonal diameter) should be the entry criterion.

Trial centres will be vascular hubs/centres able to deliver both EVAR and surveillance programmes and have an annual EVAR caseload of ≥20 cases, with audited operative mortality of <3% for EVAR (via national registry or similar standard monitoring procedures).

The trial EVAR procedures will be delivered by vascular surgeons in accredited hospitals for vascular surgery in all participating countries.

Qualitative Research to optimize recruitment

The Quintet Recruitment Intervention (QRI) will be used to identify recruitment obstacles and facilitate improvements to the recruitment process. QRI semi-structured interviews, with individuals involved in screening and presenting WARRIORS to patients, will take place across all sites (n=3-5 per site). Interviews with patients who decline randomisation will also be used to explore the reasons for not taking part in the trial. Interviews will be recorded digitally and analysed following the conventions of thematic and the constant comparison approach. Summaries of anonymised findings will be presented to WARRIORS principal investigators and to the trial management groups in each country, including supporting evidence to describe factors hindering recruitment. A potential plan of action to improve recruitment will be proposed to facilitate decision making and define responsibilities for implementation.

Screening and pre-randomisation evaluations

Participants will have a known AAA with diameter between 4.0 cm and 5.4 cm based on ultrasonography. Potential participants for the trial will have a CTA examination of the aorta, iliac and femoral arteries to assess inclusion and exclusion criteria (morphological eligibility for EVAR and presence of proximal aneurysms) unless a CTA has been completed within the previous 6 months. The baseline questionnaires for quality f life and anxiety should be administered before the eligibility assessment CTA. Women also will be assessed for Rockwood frailty score. There is no test required before the participant enters the trial. Potential participants will be screened to determine whether they meet all the inclusion criteria and none of the exclusion criteria listed for the trial. Sites will be asked to capture patient initials of each identified patient and to record the reasons for ineligibility. Women who are ineligible for the trial can opt for follow up in the associated registry.

Potential participants will be given information on the trial by local research staff when appropriate. They will be given a copy of the patient information sheet (PIS) and informed consent form (IC.F). Translations in local languages will be available, as appropriate. Patients will be given at least 24 hours to read the PIS and consider their participation.

There will be an infographic or video explanation of the trial and a decision aid which has been developed specifically for this trial.

The consent may only take place once all the above procedures are completed.

Randomization and Blinding

Randomization: 1112 women with small AAA will be randomized (1:1). Randomization will be carried out using a web-based randomization and Electronic Data Capture (EDC) system, called OpenClinica and women will be allocated to treatment using a variable block randomization schedule, stratified by country, age (≤75; >75 years) and aneurysm diameter (4.0-4.9; ≥5.0 cm) This will be generated by computer algorithm and released after checking patient eligibility and written consent.

Blinding: For ethical and practical reasons, patients and clinicians cannot be blinded to treatment allocation. However, endpoints will be adjudicated by an expert panel (PROBE study - Prospective Randomized Open, Blinded End-point).

Follow-up

Follow up visits will take place at each of the sites in a clinical examination room for interview, examination, and required questionnaires to be completed. Each study visit will be expected to take less than one hour including rest periods for the subject. For patients in the early EVAR group, follow up visits are likely to be preceded by imaging by Duplex or CT scan, to check continuing endograft exclusion of the AAA. Follow up for quality of life and anxiety questionnaires may be conducted by telephone or video conferencing, which should precede the follow up imaging study, at 1, 3 and 5 years after randomization. Data for aneurysm or other cardiovascular event treatments at hospitals not participating in the study will be collected from routine national health data sets (such as MHS Digital for English patients or Medicare in the USA).

Data will be collected on electronic case report forms using a study database hosted at Imperial College London.

INTERVENTION - Endovascular aneurysm repair (EVAR)

The purpose of EVAR is to exclude the AAA from the circulation and therefore avoid the risk of future aneurysm rupture. Many different endografts are licensed and available. Newly approved devices will be added and any advances in technology tracked. The sizing of the aorta and planning of the operation should be conducted on a 3D workstation as standard.

A protocol for pre-operative care will be recommended and include pre-operative cardiac and anaesthetic assessments and prehabilitation advice based on the 2021 guidelines from the British Geriatric Society (https://www.bgs.org.uk/cpocfrailty). This includes advice about smoking cessation, alcohol, medication adherence (e.g. antihypertensives, statin as tolerated, antiplatelet) and exercise [16,17]. Post-operatively, the recommended care will be according to European Society of Vascular Surgery 2024 guidelines. All patients (early intervention and surveillance) also should be on medications to minimise cardiovascular risk (assuming them to be in a high-risk category, with management of smoking cessation, lipid levels etc according to European Society of Cardiology guidelines.

The procedure may be performed under general, local, or regional anesthesia.

The purpose of the intervention is to reline the aorta and exclude the aneurysm from the circulation, to prevent further expansion and eventual rupture. With exclusion of the AAA from the circulation, the aneurysm sac should cease growth or decrease in diameter. Specifically in this trial the intervention will be performed when the aneurysm is between 4.0-5.4cm in size.

A strict protocol for the technical aspects of EVAR will not be given since practice around the world differs and patient differences necessitate a range of approaches. However, compliance with best practice guidelines for endovascular aortic aneurysm repair will be an expectation:

* Clinical practice guidelines EVAR: https://www.jvir.org/article/S1051-0443(10)00761-X/pdf
* Clinical practice guidelines AAA: https://www.esvs.org/wp-content/uploads/2018/12/Wanhainen-A-et-al-ESVS-AAA-GL-2019-epublished-041218.pdf
* Clinical practice guidelines AAA: https://www.jvascsurg.org/article/S0741-5214(17)32369-8/fulltext
* Manufacturers' Instructions for Use

The procedure will take place in an operating theatre environment with mobile or fixed X-Ray imaging capabilities as per local standard operating procedures. Stent graft follow-up will take place at the institution where the index procedure was performed.

There are standards outlined for a dedicated EVAR Facility. These will be used as the gold standard in this study and provided to all participating units. For specifications please see: https://www.vascularsociety.org.uk/_userfiles/pages/files/Document%20Library/mhra_8pp_leaflet_amended_more_pages_web_version.pdf

Before the procedure, pre-operative CT imaging assessment will be performed and assessed for suitability for EVAR and must meet the minimum specifications set by the Cor Laboratory. The EVAR procedure will be performed based on local assessment of the pre-operative CT scan: these will be sent to the core laboratory for independent adjudication. The participant must be suitable for EVAR using any approved device within the manufacturer's instructions for use. The sizing and planning will take place on a dedicate 3D workstation.

Before EVAR, patients will be managed according to country-specific criteria and undergo full pre-operative assessment. Each participant will be seen in the pre-operative assessment clinic with provision of participant information and supporting materials.

Pre-operative cardiac investigations will vary from country to country but at minimum should include an ECG and chest X-ray.

Any further investigations will be ordered and treatment of conditions that might cause adverse outcomes during any operative procedure or delay recovery will be undertaken at the discretion of the treating team.

Prehabilitation advice will be recommended, based on guidelines from the British Geriatric Society.

Each patient will be consented for the EVAR procedure to ensure the inclusion of EVAR competent centres with excellent safety records..

The procedure may be performed under general, regional, or local anaesthetic. Access to the arterial system will be via the common femoral artery either using a percutaneous approach (closed with any of the available closure devices) or after surgical cut down and control of the artery.

Adjuncts to facilitate delivery of the EVAR device for participants with small iliac arteries, may include:

Construction of a surgical conduit surgically to facilitate access.

Balloon angioplasty and stenting of iliac arteries

Construction of an ilio-femoral bypass

Femoral or iliac endarterectomy +/- patch plasty

Femoral or iliac patch plasty alone

The stent graft will be selected based on size measurements on the pre-operative CT scan. Each centre should only use the endografts with which they are familiar and use these within the manufacturer's IFU. A suitable oversizing of the graft as suggested by the instructions for use of the graft will be used.

Planned adjunct procedures may include:

Endoanchor or endosuture placement

Licensed branched iliac device

Licensed fusion imaging software

When considering the landing zone of the stent, the clinician will plan to land the stent in the healthy parallel neck of the aorta just below the renal arteries, consistent with the necessary landing zone requirements of the chosen endograft. Balloon moulding will be considered if appropriate following stent graft implantation.

Distally the stent will may be landed in the common iliac artery or into the external iliac artery with management of the internal iliac artery.

At the end of the procedure post-stent intra-arterial digital subtraction quality control angiogram images will be obtained. Further imaging such as rotational CT analysis will be performed at the discretion of the investigator.

Unless expected to resolve by the initial post-operative scan, in the presence of any type 1 or 3 endoleak the operating team will undertake further procedures to attempt to rectify the endoleak based on local practice and equipment provision.

Any further adjunct procedures to treat endoleak will be placed in accordance with their instructions for use. Adjunct procedures may include one or more of (but will not be limited to):

Repeat balloon moulding

Aortic extension cuff

Placement of a Palmaz (Cordis) balloon-expandable stent

Iliac extension cuff

Endoanchor placement

Chimney graft placement in the visceral/renal vessels

Post-operative care will conform to European Society of Vascular Surgery 2024 guidelines. The Enhanced Recovery After Surgery guidelines approved by the Society for Vascular Surgery will be circulated to all sites.

The participant will stay as an inpatient for standard post-operative monitoring and recovery, before being discharged. Recovery and discharge arrangements will vary from site to site and should follow standard of care pathways at that site.

After discharge from the hospital after EVAR, patients will attend for CT/MRI scan at between 3 and 12-weeks, which is clinically necessary to assess the placement of the stent. Participants will attend for subsequent clinical and imaging (either with ultrasound or CT scanning) for stent graft monitoring as directed by local follow up arrangements and the trial follow up protocol.

During the trial period modifications of the procedure and devices will be expected as new technology if developed. The procedural/device modifications will be tracked to ensure that the results of the outcomes from EVAR are not affected positively or negatively, leading to errors in the trial conclusions.

STANDARD MANAGEMENT - Surveillance with ultrasound (or other imaging) surveillance with delayed repair for rupture or aneurysm diameter reaching 5.5 cm threshold

All women will be monitored for AAA growth. Ultrasonographic surveillance is the preferred method since it is non-invasive, whilst being highly sensitive and specific, although in some countries (e.g. USA), CT, including non-contrast CT, may be used for surveillance. For AAA between 4.0-4.4 cm diameter, annual surveillance can be recommended, increasing to every 6 months for AAA of 4.5 cm diameter or greater or according to current local practice and standard operating procedures. For ultrasound surveillance, the anterior-posterior diameter should be measured in the longitudinal plane, since this is more repeatable than the transverse diameter. Calliper placement for measurements should be consistent at each surveillance visit. Outer-to-outer diameter measurements are preferred, but where sonographers are trained to measure either leading edge to leading edge or inner-to-inner diameters, these methods should be used and documented. When CT imaging is used for surveillance the centreline orthogonal diameter should be measured. When the diameter exceeds 5.4 cm the participant should have a prompt (target within 2 weeks) consultation with a vascular surgeon consideration of AAA repair by which ever method is recommended by the local team. The operation CRF should be completed, and the participant will then enter routine clinical follow up.

If there is any suspicion of AAA rupture, the patient must be admitted immediately as an emergency, preferably to a vascular surgeon the site where the patient has been followed up.

If there is a suspicion of impending rupture, with symptoms of back or abdominal pain referable to the aneurysm, further investigations should be performed, and consideration given to early elective repair. Thromboembolic evens referable to the aneurysm are also an indication for consideration of early elective (urgent) repair. (These conditions are known as symptomatic AAA).

All randomized patients will be offered smoking cessation advice and adjunct therapies as well as best medical therapy, including statins with a cardiologist-guided protocol (European Society of Cardiology guidelines for the high-risk category). This protocol will include and exercise, blood pressure, body weight and LDL-cholesterol targets and good diabetic control where relevant[. All patients will receive advice about exercise and physical activity. These measures will be conducted using patient-facing educational resources and through communication with their General/Family Practitioner.

Permanent Discontinuation of Study Intervention and Withdrawal from Study

Permanent discontinuation of study intervention

Participants may discontinue study intervention for the following reasons:

At the request of the participant.

Adverse event/ Serious Adverse Event

If the investigator considers that a participant's health will be compromised due to adverse events or concomitant illness that develop after entering the study.

Withdrawal from Study

Withdrawal from the study refers to discontinuation of study intervention and study procedures and can occur for the following reasons:

Participant decision

Loss to follow-up

Procedures for Withdrawal from Study

If a subject withdraws prematurely the reason for withdrawal will be recorded in the CRF/eCRF and medical records. All study visits up to the point of any planned withdrawal will be completed.

SAFETY REPORTING

Adverse Event (AE)

An AE is any untoward medical occurrence in a SAFETY REPORTING

Adverse Event (AE)

An AE is any untoward medical occurrence in a patient or clinical trial participant. An AE can therefore be any unfavourable and unintended sign (including an abnormal laboratory finding), symptom, whether or not considered related to the trial protocol.

Adverse Event recording

Adverse events will be assessed at each study visit. The following will be assessed for all adverse events:

date of onset

description of event

frequency

severity

causality

outcomes

action taken.

For the purposes of the study, AEs will be followed up according to local practice until the event has stabilised or resolved, or the follow-up visit, whichever is the sooner.

Adverse events that are not serious adverse events will only be recorded on adverse event forms if the adverse event either occurs within 90 days of the index AAA repair or is aortic related. The following will be noted as aortic related events:

Any events within 30 days of index repair

Access vessel dissection or rupture

Buttock claudication

Endoleak

Graft kinking (clinically significant)

Graft migration of >5mm

Graft limb thrombosis/stenosis/occlusion

Limb ischaemia or toe amputation

New onset claudication

Pseudo-aneurysm at graft insertion site

Surgical site infection

All SAEs will be recorded throughout the study.

Severity of Adverse Events

The assessment of severity will conform to the following definitions:

Mild: Awareness of event but easily tolerated

Moderate: Discomfort enough to cause some interference with usual activity

Severe: Inability to carry out usual activity

Causality of Adverse Events

The assessment of causality will conform to the following definitions:

Unrelated: No evidence of any causal relationship

Unlikely: There is little evidence to suggest there is a causal relationship and there is another reasonable explanation for the event (e.g. the participant's clinical condition, other concomitant treatment).

Possible: There is some evidence to suggest a causal relationship. However, the influence of other factors may have contributed to the event (e.g. the participant's clinical condition, other concomitant treatments).

Probable: There is evidence to suggest a causal relationship and the influence of other factors is unlikely.

Definite: There is clear evidence to suggest a causal relationship and other possible contributing factors can be ruled out.

Serious Adverse Events (SAE)

Definition of SAE

An SAE is defined as any event that

Results in death;

Is life-threatening (eg aortic rupture)*;

Requires hospitalisation or prolongation of existing inpatient's hospitalisation (eg graft infection or conversion to open repair)**;

Results in persistent or significant disability or incapacity (e.g. major limb amputation);

* "Life-threatening" in the definition of "serious" refers to an event in which the participant was at risk of death at the time of the event; it does not refer to an event which hypothetically might have caused death if it were more severe.

** "Hospitalisation" means any unexpected admission to a hospital department. It does not usually apply to scheduled admissions that were planned before study inclusion or visits to casualty (without admission).

ELIGIBILITY:
Inclusion Criteria:

* female sex
* age ≥50 years
* infra-renal abdominal aortic aneurysm with a maximum infrarenal aortic anterior-posterior diameter 4.0-5.4 cm, aneurysm, measured on ultrasonography or the centreline orthogonal diameter on Computed Tomography (CT) scan when this is the discovery imaging mode,
* Local assessment that arterial morphology is suitable for EVAR within manufacturer's IFU for any licensed infrarenal endograft, including those with concomitant common iliac aneurysm(s), provided the device is landed in the iliac arteries, without coverage of patent internal iliac arteries.
* Rockwood frailty score <7.

Exclusion Criteria:

* Male sex
* aneurysm of the infrarenal aorta of <4.0 or >5.4cm
* infrarenal aneurysm not meeting IFU for any specific licensed endograft for standard EVAR
* inability to give informed consent
* previous abdominal aortic surgery
* age <50 years
* concomitant thoracic aortic aneurysm of >4.0cm diameter
* excessive frailty (Rockwood frailty score 7 or more)
* life expectancy <2 years (in the opinion of the site principal investigator)
* severe contrast allergy not amenable to steroid/antihistamine pretreatment (e.g., anaphylaxis)
* those considered unlikely to comply with follow-up
* concomitant common iliac artery aneurysm unless: a) the arterial morphology is within the IFU for standard infrarenal EVAR; or b) the arterial morphology is suitable for a licensed iliac branch device; or c) the internal iliac artery is occluded and the stent limb can be landed in the external iliac artery without embolization of the internal iliac artery.

There will be no patient excluded as a result of geographical location, disability, gender, marriage and civil partnership status, ethnicity, religion or belief, sexual orientation, socioeconomic status or access to health or social care.

Min Age: 50 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 1112 (Estimated)
Dates: Start 2025-07-01 (Estimated); Primary Completion 2033-10-31 (Estimated); Study Completion 2034-04-30 (Estimated)

PRIMARY OUTCOMES:
Aneurysm-related mortality and rupture | To at least 5 years
  Death caused by the aneurysm or its treatment and non-fatal rupture. Aneurysm-related mortality will include any death within 30 days of AAA repair, death in hospital at beyond 30 days for the index admission for AAA repair and at the same time-points after reinterventions following the index AAA repair, and death from repair or rupture of a supra-renal or iliac aneurysm.

SECONDARY OUTCOMES:
Quality-Adjusted Life Years | 5 years
  Quality of life (from EuroQol 5D-5L questionnaire,, scale 0 to 1, with 1 being best quality of life)) integrated with respect to overall survival.

OTHER OUTCOMES:
Anxiety | 5 years
  Anxiety assessed from Hospital Anxiety & Depression Scale (HADS, 0-21, lowes tscores mean most anxious)) questionnaire
Major Adverse Cardiovascular events | 5 years
  Myocardial infarction, stroke and lower limb amputation
Hospital costs | 5 years
  For aneurysm treatment, (both in-patient and out-patient)
cost-effectiveness | 5 years
  combining data for quality of life (using EuroQol 5D-5L as in outcome 2 above) and hospital treatment costs
loss of eligibility for EVAR | 5 years
  changes in aortic morphologyc, since screening CT scan, so that standard infrarenal EVAR is not recommended in surveillance patients who have not undergone aneurysm repair. This will be determined by the core laboratorynfor CT scans.

CONTACTS AND LOCATIONS:
Overall Officials: Alison Halliday, FRCS, Study Chair — University of London

IPD SHARING:
Plan to Share IPD: Yes
only pseudo-anonymised data will be shared requests to be adjudicated by central trial management committee
Supporting Information: Study Protocol, SAP, ICF
Time Frame: Available on the trial website now
Access Criteria: Website
URL: https://www.imperial.ac.uk/department-surgery-cancer/research/surgery/clinical-trials/international-warriors-trial/